CLINICAL TRIAL: NCT00560716
Title: A Phase I Pharmacologic Study of CYC116, an Oral Aurora Kinase Inhibitor, in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYC116-06-01; NCT00530465 (obsolete NCT alias)
Record Dates: First submitted 2007-11-16; First posted 2007-11-20 (Estimated); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — 4-methyl-5-(2-(4-morpholinophenylamino)pyrimidin-4-yl)thiazol-2-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CYC116 (Experimental): CYC116 dose escalation first-in-human evaluation
  Interventions: Drug: CYC116

INTERVENTIONS:
Drug: CYC116 — Dose escalation of CYC116
  Other Names: Aurora kinase inhibitor

SUMMARY:
This is a phase I study of an investigational cancer drug, CYC116, in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Phase I study of an investigational cancer drug, CYC116, an Aurora kinase inhibitor, in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Incurable advanced solid tumors that did not respond to conventional therapy or for which no effective therapy exists
* Age >=18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy ≥ 3 months
* Evaluable disease
* Adequate bone marrow function
* Adequate renal function
* Adequate liver function
* At least 3 weeks from prior systemic treatments including investigational anti-cancer therapy, radiation therapy; and have recovered from prior toxicities
* Able to swallow capsules
* At least 3 weeks from major surgery
* Agree to practice effective contraception

Exclusion Criteria:

* Previously untreated CNS metastasis or progressive CNS metastasis documented by MRI scan performed at 4 weeks or longer after the last treatment for CNS metastasis
* Currently receiving radiotherapy, biological therapy, or any other investigational agents
* Uncontrolled intercurrent illness
* Pregnant or lactating women
* Known to be HIV-positive
* Known active hepatitis B and/or hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-06; Primary Completion 2009-01 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | over the course of study
  Safety and tolerability; SAEs and AEs

CONTACTS AND LOCATIONS:
Overall Officials: Judy H Chiao, MD, Study Director — Cyclacel Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No